CLINICAL TRIAL: NCT06255951
Title: This is a Single-center, Two-sequence, Open-label, Two-cycle Drug-drug Interaction (DDI) Study in Healthy Subjects. To Evaluate the Effects of Itraconazole Capsules, a Strong Inhibitor of CYP3A4, and Rifampicin Capsules, a Strong Inducer, on the Pharmacokinetics of TY-9591 Tablets After a Single Oral Dose
Brief Title: Studies Evaluating the Effects of Itraconazole or Rifampicin on the Pharmacokinetics of TY-9591 Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TYK Medicines, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TYKM1601105
Record Dates: First submitted 2024-01-17; First posted 2024-02-13 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: NSCLC
MeSH Terms: interventions — Itraconazole; Rifampin

STUDY DESIGN:
Intervention Model Description: PartA is the itraconazole study sequence,PartB was the rifampin study sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Itraconazole (Experimental): Itraconazole
  Interventions: Drug: Itraconazole
- Rifampicin (Experimental): Rifampicin
  Interventions: Drug: Rifampicin

INTERVENTIONS:
Drug: Itraconazole — The study was divided into two sequences with a planned enrollment of 48 healthy adult subjects (24 in each sequence). PartA was the itraconazole study sequence, which was used to study the effect of itraconazole on the pharmacokinetic characteristics of TY-9591 tablets after multiple doses.
  Arms: Itraconazole
Drug: Rifampicin — The study was divided into two sequences with a planned enrollment of 48 healthy adult subjects (24 in each sequence). PartB was the rifampin study sequence, which investigated the effect of multiple doses of rifampin on the pharmacokinetic profile of TY-9591 tablets.
  Arms: Rifampicin

SUMMARY:
Studies evaluating the effects of itraconazole or rifampicin on the pharmacokinetics of TY-9591 tablets in healthy subjects

DETAILED DESCRIPTION:
To evaluate the pharmacokinetics of TY-9591 tablets in healthy Chinese subjects after a single oral administration. To evaluate the effects of itraconazole/rifampicin on the pharmacokinetics of TY-9591 and its metabolites D1 and D2 after oral administration of TY-9591 tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female healthy adult subjects aged 18-45 years old (inclusive), in which male or female accounted for no less than 1/4 of the total number of subjects in each sequence.
2. Body mass index (BMI) between 19.0 and 26.0 kg/m2 [BMI= weight (kg)/ height 2 (m2)] (including boundary values).
3. Participants (including male participants) were infertile themselves, or agreed to use highly effective nonpharmacologic contraceptive methods or abstain completely from sex for 6 months after the last dose of self-medication.
4. Subjects voluntarily participated and signed an informed consent form.
5. Subjects had good communication with investigators and were able to complete the trial in accordance with the protocol.

Exclusion Criteria:

1. Those with clinically significant abnormalities in physical examination, vital signs, routine laboratory tests (blood routine, urine routine, blood biochemistry, coagulation function), 12-lead electrocardiogram, ophthalmic examination, abdominal color Doppler ultrasound (liver, bile duct, pancreas, spleen, kidney), etc.
2. Persons with one or more positive results of human immunodeficiency virus (HIV) antibody, hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV) antibody, or treponema pallidum antibody (Anti-TP).
3. smokers with an average of more than 10 cigarettes per day in the previous 3 months or habitual users of nicotine products who could not quit during the study.
4. Heavy drinking or regular drinking in the 3 months before the screening period, i.e. drinking more than 14 units of alcohol per week (1 unit =360 mL of beer or 45 mL of 40% spirits or 150 mL of wine); Or alcohol breath test results on admission > 0.0 mg/100 mL and those who could not abstain from alcohol during the experiment.
5. those who consumed excessive amounts of tea, coffee, and/or caffeinated beverages (average > 8 cups/day, 250 mL/cup) in the 3 months before the screening period, and those who could not stop using them during the study period.
6. those who took dragon fruit, mango, grapefruit, chocolate, any food or beverage containing caffeine, diet rich in xanthine, and other special diets affecting drug absorption, distribution, metabolism, and excretion within 7 days before taking the drug.
7. Use of any drugs that inhibit or induce the liver CYP3A4 enzyme (see Appendix II), herbs, or foods containing herbal ingredients within 30 days before the screening period.
8. taking any medicine (including Chinese herbal medicine and health supplements) within 14 days before taking the test drug.
9. enrollment in any drug clinical trial within 3 months before the screening period.
10. Subjects who may not be able to complete the study for other reasons or who are considered unsuitable for the study by the investigators.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentrations (Cmax) of TY-9591 and its metabolites D1 and D2 | through study completion,an average of 6 months
  Peak plasma concentrations (Cmax) of TY-9591 and its metabolites D1 and D2
Area under the concentration-time curve from 0 to the last quantifiable time point after dose administration (AUC0-t) | through study completion,an average of 6 months
  Area under the concentration-time curve from 0 to the last quantifiable time point after dose administration (AUC0-t)
Area under the concentration-time curve from 0 to infinity (AUC0-inf), as data permit | through study completion,an average of 6 months
  Area under the concentration-time curve from 0 to infinity (AUC0-inf), as data permit

SECONDARY OUTCOMES:
Time to peak concentration (Tmax) of TY-9591 and its metabolites D1 and D2 | through study completion,an average of 6 months
  Time to peak concentration (Tmax) of TY-9591 and its metabolites D1 and D2
The half-life of elimination phase (t1/2) of TY-9591 and its metabolites D1 and D2 | through study completion,an average of 6 months
  The half-life of elimination phase (t1/2) of TY-9591 and its metabolites D1 and D2
elimination rate constant (λz) of TY-9591 and its metabolites D1 and D2 | through study completion,an average of 6 months
  elimination rate constant (λz) of TY-9591 and its metabolites D1 and D2
apparent clearance rate (CL/F) of TY-9591 and its metabolites D1 and D2 | through study completion,an average of 6 months
  apparent clearance rate (CL/F) of TY-9591 and its metabolites D1 and D2
apparent volume of distribution (Vd/F) of TY-9591 and its metabolites D1 and D2 | through study completion,an average of 6 months
  apparent volume of distribution (Vd/F) of TY-9591 and its metabolites D1 and D2
mean retention time (MRT) of TY-9591 and its metabolites D1 and D2 | through study completion,an average of 6 months
  mean retention time (MRT) of TY-9591 and its metabolites D1 and D2
Cmax ratio of metabolites to original drug | through study completion,an average of 6 months
  Cmax ratio of metabolites to original drug
AUC ratio of metabolites to original drug | through study completion,an average of 6 months
  AUC ratio of metabolites to original drug

CONTACTS AND LOCATIONS:
Overall Officials: yali liu, Principal Investigator — Investigator
Locations (1):
- Yali Liu, Guangdong, Shantou, China

IPD SHARING:
Plan to Share IPD: No